CLINICAL TRIAL: NCT04248569
Title: A Pilot Study of a DNAJB1-PRKACA Fusion Kinase Peptide Vaccine Combined With Nivolumab and Ipilimumab for Patients With Fibrolamellar Hepatocellular Carcinoma
Brief Title: DNAJB1-PRKACA Fusion Kinase Peptide Vaccine Combined With Nivolumab and Ipilimumab for Patients With Fibrolamellar Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Fibrolamellar Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J19140; IRB00222681 (Other: Johns Hopkins Medicine Institutional Review Board)
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Fibrolamellar Hepatocellular Carcinoma (FLC)
Keywords: DNAJB1-PRKACA Peptide Vaccine; Nivolumab; Ipilimumab; Anti-PD-1 (receptor blocking antibody); Anti-CTLA-4 (receptor blocking antibody); Neoantigen Vaccines; Cancer Vaccines; Immunotherapy; Fibrolamellar Hepatocellular Cancer (FLC)
MeSH Terms: conditions — Fibrolamellar hepatocellular carcinoma | interventions — poly ICLC; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DNAJB1-PRKACA peptide vaccine, Nivolumab, and Ipilimumab (Experimental): Cohort A: Patients with FLC cancer with no prior checkpoint inhibitor treatment. Cohort B: Patients with FLC cancer with prior checkpoint inhibitor treatment. Cohort C: Patients with non-FLC cancer (solid tumors) with prior checkpoint inhibitor treatment eligible.
  Interventions: Drug: DNAJB1-PRKACA peptide vaccine; Drug: Nivolumab; Drug: Ipilimumab
- R- Enrollment: DNAJB1-PRKACA peptide vaccine, Nivolumab, and Ipilimumab (Experimental): Re-enrolling patients: Patients previously treated with the vaccine targeting the DNAJB1-PRKACA fusion kinase in combination with nivolumab and ipilimumab, who, in the opinion of the principal investigator, had clinical or radiological benefits. Re-enrolling patients who come off treatment ≤ 12 months from last dose may resume therapy at the study timepoint that they stopped study therapy. Patients who came off study therapy > 12 months of last dose (i.e. to pursue alternative therapies (for example, surgical debulking), or after completion of the 2 years of study therapy), may restart study therapy at C1D1. In both cases, if the investigator assesses a drug-related toxicity to be related to anti-CTLA4 (ie. not anti-PD(L)1) therapy, patients can be enrolled in the study with nivolumab plus FLC peptide vaccine only.
  Interventions: Drug: DNAJB1-PRKACA peptide vaccine; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: DNAJB1-PRKACA peptide vaccine — 1. DNAJB1-PRKACA peptide vaccine: Day 1, 8, 15 of cycle 1 and on Day 1 of cycle 2, 3 and 4 (priming phase). Boost vaccinations: every 3 cycles beginning C5D1.
  2. Drug: 0.3 mg DNAJB1-PRKACA peptide vaccine + 0.5mg Poly-ICLC
  Other Names: Hiltonol® (Poly-ICLC)
Drug: Nivolumab — 1. Nivolumab 3mg/kg will be administered as a 30 minute IV infusion (-10/+15min) on Day 1 of Cycle 1-4 during the priming phase. Boost/maintenance vaccinations will be administered as a flat dose of 480mg every 4 weeks starting on Day 1 of Cycle 5.
  2. Drug: 3mg/kg and 480mg IV
  Other Names: OPDIVO
Drug: Ipilimumab — 1. Ipilimumab (1 mg/kg) will be administered as a 30 minute IV infusion (-10/+15min) on Day 1 of Cycles 1, 2, 3 and 4 of the study, every 3 weeks of the priming phase.
  2. Drug: 1mg/kg IV
  Other Names: YERVOY®

SUMMARY:
The primary objective of the trial is the safety and tolerability of administering a vaccine targeting the DNAJB1-PRKACA fusion kinase, in combination with nivolumab and ipilimumab in patients with unresectable or metastatic FLC and with non-FLC solid tumors and to assess the T-cell response.

ELIGIBILITY:
Inclusion Criteria for Cohort A, B and C:

* Cohort A and B: Must have histologically confirmed FLC (fibrolamellar hepatocellular cancer) that is metastatic or unresectable.
* Cohort C: Patients with histologically proven metastatic or unresectable DNAJB1-PRKACA fusion transcript positive solid tumor malignancies, non-FLC solid tumors.
* Cohort A and B: Age > 12 years. Note: Subjects age > 12 years but <18 are eligible to enroll only after 6 adult patients have enrolled on the study.
* Cohort A and B: Patients < 18 years old must have a body weight ≥40 kg.
* Cohort C: Patients must be Age ≥ 18 years.

All Cohorts:

* Presence of DNAJB1-PRKACA fusion transcript, assessed by RNA-sequencing, DNA-sequencing, or in situ hybridization in the archival tissue.
* ECOG performance status of ≤2 (Karnofsky ≥60%)
* Patients must have adequate liver, kidney and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Patients must have measurable disease per RECIST 1.1.
* Must be willing to provide tissue and blood samples for mandatory translational research.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Men must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria for Cohorts A, B and C:

* Cohort A and C: Patients with a history of prior treatment with checkpoint inhibitors, such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40, anti-CTLA-4, or anti-LAG-3 antibodies. NOTE: Prior therapy with interferon-alpha is allowed.
* Cohort B: Participants a with history of unacceptable, life-threatening toxicity related to prior immune therapy (eg, anti-CTLA-4 or anti-PD-1/PD-L1 treatment, any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (eg, hormone replacement after endocrinopathy).

All Cohorts:

* Have had chemotherapy or other systemic therapy or radiotherapy, as follows:

  * Have had chemotherapy, biological cancer therapy, or radiation 14 days prior to the first dose of study drug.
  * Have had surgery within 28 days of dosing of investigational agent, excluding minor procedures (dental work, skin biopsy, etc.), celiac plexus block, and biliary stent placement.
  * Have received other approved or investigational agents or device within 28 days of the first dose of study drug.
  * Have not recovered from acute adverse events to grade ≤1 or baseline due to agents administered.
* Have received any non-oncology live vaccine therapy used for prevention of infectious diseases within 28 days of study treatment
* Known sensitivity to or history of allergic reactions to investigational drug (s).
* Hypersensitivity reaction to any monoclonal antibody.
* Has active autoimmune disease that has required systemic treatment in the past 2 years, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Presence of any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft. Patients with a history of allogeneic hematopoeitic stem cell transplant will be excluded.
* Has a diagnosis of immunodeficiency.
* Systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of study drug administration.
* Symptomatic interstitial lung disease.
* Has a pulse oximetry of <92% on room air or is on supplemental home oxygen.
* Active or untreated brain metastases or leptomeningeal metastases.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Are pregnant or breastfeeding.
* Infection with HIV or hepatitis B or C.
* Have had evidence of active or acute diverticulitis, intra-abdominal abscess, or GI obstruction.
* Unwilling or unable to follow the study schedule for any reason.
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Any illicit drugs or other substance abuse.
* Clinically meaningful ascites.

Inclusion Criteria for Re-Enrolling Patients:

* Patients previously treated with the vaccine targeting the DNAJB1-PRKACA fusion kinase in combination with nivolumab and ipilimumab, who, in the opinion of the principal investigator, had clinical or radiological benefits.
* Patients < 18 years old must have a body weight ≥40 kg.
* ECOG performance status of ≤2 (Karnofsky ≥60%, see Appendix A).
* Patients must have adequate liver, kidney and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Patients must have measurable disease per RECIST 1.1.
* Willingness to provide tissue and blood samples for mandatory translational research.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Men must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria for Re-Enrolling Patients:

* Participants with a history of prior unacceptable and/or life-threatening toxicities.
* Patients who have had chemotherapy or other systemic therapy or radiotherapy, as follows:

  * Patients who have had chemotherapy, biological cancer therapy, or radiation 14 days prior to the first dose of study drug.
  * Patients who have had surgery within 28 days of dosing of investigational agent, excluding minor procedures (dental work, skin biopsy, etc.), celiac plexus block, and biliary stent placement.
  * Patients who have received other approved or investigational agents or device within 28 days of the first dose of study drug.
  * Patients who have not recovered from acute adverse events to grade ≤1 or baseline due to agents administered, with exception of alopecia or stable neuropathy, unless approved by the IND Sponsor.
* Patients who have received any non-oncology live vaccine therapy used for prevention of infectious diseases within 28 days of study treatment.
* Known sensitivity to or history of allergic reactions to investigational drug (s).
* Hypersensitivity reaction to any monoclonal antibody.
* Has active autoimmune disease that has required systemic treatment in the past 2 years, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Has active autoimmune disease that has required systemic treatment in the past 2 years, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Presence of any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft. Patients with a history of allogeneic hematopoeitic stem cell transplant will be excluded.
* Has a diagnosis of immunodeficiency.
* Systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of study drug administration.
* Symptomatic interstitial lung disease.
* Has a pulse oximetry of <92% on room air or is on supplemental home oxygen.
* Active or untreated brain metastases or leptomeningeal metastases.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Are pregnant or breastfeeding.
* Infection with HIV or hepatitis B or C.
* Have had evidence of active or acute diverticulitis, intra-abdominal abscess, or GI obstruction.
* Unwilling or unable to follow the study schedule for any reason.
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Any illicit drugs or other substance abuse.
* Clinically meaningful ascites.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2034-03-01 (Estimated)

PRIMARY OUTCOMES:
All Cohorts: Number of participants experiencing study drug-related toxicities | 4 years
  Number of participants experiencing study drug-related adverse events Grade 3 or higher as defined by CTCAE v5.0
All Cohorts: Fold change in interferon-producing DNAJB1-PRKACA-specific CD4 and CD8 T cells at 10 weeks | Baseline and 10 weeks
  Evaluated by the fold change in interferon-producing DNAJB1-PRKACA-specific CD8 cells after vaccination at 10 weeks compare to pre-vaccination baseline.
Cohort A only: Progression-free survival (PFS) | 6 months
  PFS at 6 months, will be estimated as the proportion of subjects who remain alive and free of disease progression at 6 months from the start of treatment. Disease progression will be determined using RECIST 1.1 criteria. The proportion of subjects achieving PFS at 6 months will be estimated using the Kaplan-Meier method, and the corresponding 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 4 years
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Duration of response (DoR) | 4 years
  Number of weeks from the start date of PR or CR (whichever response is recorded first) and subsequently confirmed to the first date of disease progression or death is documented per RECIST 1.1. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions.
Disease control rate (DCR) | 4 years
  DCR is defined as the number of patients achieving a complete response (CR) or partial response (PR) and stable disease (SD) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Progression-free survival (PFS) | 4 years
  PFS is defined as number of months from the date of first treatment until first documented local progression or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Overall survival (OS) | 4 years
  OS will be measured from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yarchoan, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baretti M, Kirk AM, Ladle BH, Kamdar Z, Bendinelli KJ, Ho WJ, Adhikari S, Clark NA, Sundararaman B, Wang H, Kung HC, Hernandez J, Qi H, Shin SM, Hernandez A, Nakazawa M, Schattgen SA, Crawford JC, Furth M, Anders RA, Thoburn C, Zaidi N, Huff AL, Nauroth J, Jaffee E, Pogorelyy MV, Thomas PG, Yarchoan M. A therapeutic peptide vaccine for fibrolamellar hepatocellular carcinoma: a phase 1 trial. Nat Med. 2025 Dec;31(12):4246-4255. doi: 10.1038/s41591-025-03995-y. Epub 2025 Nov 24. PMID 41286513
- [Derived] Short SS, Kastenberg ZJ, Wei G, Bondoc A, Dasgupta R, Tiao GM, Watters E, Heaton TE, Lotakis D, La Quaglia MP, Murphy AJ, Davidoff AM, Mansfield SA, Langham MR, Lautz TB, Superina RA, Ott KC, Malek MM, Morgan KM, Kim ES, Zamora A, Lascano D, Roach J, Murphy JT, Rothstein DH, Vasudevan SA, Whitlock R, Lal DR, Hallis B, Butter A, Baertschiger RM, Lapidus-Krol E, Putra J, Tracy ER, Aldrink JH, Apfeld J, Le HD, Park KY, Rich BS, Glick RD, Fialkowski EA, Utria AF, Meyers RL, Riehle KJ. Histologic type predicts disparate outcomes in pediatric hepatocellular neoplasms: A Pediatric Surgical Oncology Research Collaborative study. Cancer. 2022 Jul 15;128(14):2786-2795. doi: 10.1002/cncr.34256. Epub 2022 May 13. PMID 35561331
- [Derived] O'Neill AF, Church AJ, Perez-Atayde AR, Shaikh R, Marcus KJ, Vakili K. Fibrolamellar carcinoma: An entity all its own. Curr Probl Cancer. 2021 Aug;45(4):100770. doi: 10.1016/j.currproblcancer.2021.100770. Epub 2021 Jul 1. PMID 34272087